CLINICAL TRIAL: NCT00382980
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Clinical Trial of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Immunization With Inactivated, Vero Cell-Culture Derived Influenza A/H5N1 Vaccine Given Alone or With Aluminum Hydroxide to Healthy Young Adults
Brief Title: Dose-Escalating Trial Using Vero Cell-culture Derived H5N1 +/- Aluminum in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-0052
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-09

CONDITIONS: Influenza
Keywords: influenza, vaccine, A/H5N1, aluminum hydroxide, Vero cell
MeSH Terms: conditions — Influenza, Human | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- 7.5- (Experimental): 7.5 mcg of vaccine without adjuvant administered on Days 0 and 28.
  Interventions: Biological: Inactivated Vero cell based whole virus influenza A/H5N1
- 45- (Experimental): 45 mcg of vaccine without adjuvant administered on Days 0 and 28.
  Interventions: Biological: Inactivated Vero cell based whole virus influenza A/H5N1
- Placebo (Placebo Comparator): Placebo administered on Days 0 and 28.
  Interventions: Drug: Placebo
- 15+ (Experimental): 15 mcg of vaccine with aluminum hydroxide adjuvant administered on Days 0 and 28.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Vero cell based whole virus influenza A/H5N1
- 7.5+ (Experimental): 7.5 mcg of vaccine with aluminum hydroxide adjuvant administered on Days 0 and 28.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Vero cell based whole virus influenza A/H5N1
- 15- (Experimental): 15 mcg of vaccine without adjuvant administered on Days 0 and 28.
  Interventions: Biological: Inactivated Vero cell based whole virus influenza A/H5N1

INTERVENTIONS:
Biological: Aluminum hydroxide — Adjuvant administered with A/H5N1 vaccine dosages 7.5 mcg and 15 mcg.
  Arms: 15+; 7.5+
Biological: Inactivated Vero cell based whole virus influenza A/H5N1 — Inactivated Vero cell-grown, whole virus, influenza A/H5N1 vaccine at dosages 7.5 mcg and 15 mcg of hemagglutinin (HA) per 0.5 mL, each dosage with and without aluminum hydroxide adjuvant; 45 mcg HA/0.5 mL without adjuvant.
  Arms: 15+; 15-; 45-; 7.5+; 7.5-
Drug: Placebo — Saline injected into the deltoid muscle. 2 identical dosages will be given approximately 28 days apart.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to compare how the body reacts to different strengths of an experimental cell culture-grown whole virus A/H5N1 flu vaccine when given with or without the addition of aluminum hydroxide adjuvant. Researchers will also look at how much antibody is made to the influenza virus hemagglutinin (HA) after subjects receive the H5N1 vaccine. Three hundred healthy adults aged 18-40 years will participate for approximately 9 months, which includes screening. Participants will receive 2 doses of vaccine or placebo injected 28 days apart. Participants will have blood samples taken up to 7 times and have 8 scheduled study visits.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, placebo-controlled, dose-ranging clinical trial of the safety, reactogenicity, and immunogenicity of intramuscular immunization with inactivated, Vero cell-culture derived influenza A/H5N1 vaccine given alone or with aluminum hydroxide to healthy young adults. The primary objectives are to determine the dose-related safety of an inactivated, cell-culture grown whole virus influenza A/H5N1 vaccine with or without aluminum hydroxide adjuvant in healthy adults; to determine the potential for aluminum hydroxide to enhance the immune response to inactivated whole virus H5N1 vaccine in healthy adults approximately 1 month following receipt of 2 doses of vaccine; and to provide information for the selection of the best dosage level for further studies. The secondary objective is to evaluate dose-related immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination. The primary endpoints are adverse event (AE) or serious adverse event (SAE) information (solicited in the clinic and via memory aids, concomitant medications, periodic targeted physical assessment, and laboratory safety evaluations in a subset of subjects); proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine (approximately Day 56); proportion of subjects in each dose group achieving a serum hemagglutination inhibition (HAI) antibody titer of greater than or equal to 40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine (approximately Day 56); geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 28 days after receipt of the second dose of vaccine; and GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 28 days after receipt of the second dose of vaccine (approximately Day 56). The secondary endpoints are GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; and GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine. Approximately 300 healthy adults, 18-40 years old inclusive, will be enrolled at up to 5 sites in the United States for up to 9 months, including the screening period. Two doses of vaccine or placebo will be injected into the deltoid muscle approximately 28 days apart. The study will be conducted in 2 stages. During Stage 1, 90 subjects will be randomized to receive saline placebo or 7.5 micrograms (with or without aluminum hydroxide), 15 micrograms (with or without aluminum hydroxide), or 45 micrograms (without aluminum hydroxide) (6 groups; N=15 per group). Blood for safety evaluations will be obtained from all subjects in the Stage 1 cohort at screening, and before and 1 week after each vaccination. Subjects in Stage 1 will receive their second vaccinations following review of available clinical and laboratory safety data by the Safety Monitoring Committee (SMC). If no dose-limiting toxicity or safety-related issues are noted during the week after administration of the first dose of vaccine during Stage 1 (based on review of clinical and laboratory safety data by the SMC), then Stage 1 subjects will receive a second vaccination. A complete Stage 1 safety report will be reviewed by the SMC prior to the enrollment of the 210 additional subjects in Stage 2 (N=50 per formulation group total). Sera for immune assessment of antigen-specific immune responses will be collected from all subjects at baseline (Day 0), 1 month after each vaccine dose, and 6 months after the second vaccine dose. This study is linked to DMID protocol 07-0022.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 Cohort

* Healthy males and females aged 18 to 40 years, inclusive;
* Females of childbearing potential must agree to practice adequate contraception for the duration of the study (not surgically sterile or Aftermenopausal for at least 1 year);
* Good health as determined by screening medical history and physical examination;
* On no medications with the exception of licensed hormonal contraceptives and vitamins;
* Willingness to comply with study procedures;
* Ability to provide informed consent;
* Availability for follow-up for 6 months after second vaccination;
* Normal screening laboratory values for total WBC, platelet count, hemoglobin, creatinine, and alanine aminotransferase (Stage 1 only).

Stage 2 Cohort

* Healthy males and non-pregnant females aged 18 to 40 years, inclusive.
* Females of childbearing potential must agree to practice adequate contraception for the duration of the study.
* Good health as determined by screening medical history and physical examination.
* Willingness to comply with study procedures.
* Ability to provide informed consent.
* Availability for follow-up for 6 months after second vaccination.

Exclusion Criteria:

Stage 1 Cohort

* Have a positive urine or serum pregnancy test in the 24 hours prior to vaccination (if female of childbearing potential) or are women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (This includes, but is not limited to, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.)
* Have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during the 7-month study period.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (but does not exclude documented placebo recipients).
* Have a known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Have a history of Guillain Barre Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Stage 2 Cohort

* Have a positive urine or serum pregnancy test prior to vaccination (if female of childbearing potential) or are women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy. Have long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, Bi-polar disease or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Are receiving psychiatric drugs*. Subjects who are receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.

  * aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, molindone, thiothixene, pimozide, fluphenazine, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (This includes, but is not limited to, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.)
* Have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during the 7-month study period.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (but does not exclude documented placebo recipients).
* Have a known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Have a history of Guillain Barre Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) or serious adverse event (SAE) information (solicited in the clinic and via memory aids, concomitant medications, periodic targeted physical assessment, and laboratory safety evaluations for a subset of subjects. | Duration of study.
Proportion of subjects in each dose group achieving a serum neutralizing antibody titer of greater than or equal to 40 against the influenza A/H5N1 virus. | 28 days after receipt of the 2nd dose of vaccine, approximately Day 56.
Proportion of subjects in each dose group achieving a serum hemagglutination inhibition (HAI) antibody titer of greater than or equal to 40 against the influenza A/H5N1 virus. | 28 days after receipt of the 2nd dose of vaccine, approximately Day 56.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group. | 28 days after receipt of the 2nd dose of vaccine, approximately Day 56.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in serum HAI antibody titers in each group. | 28 days after receipt of the 2nd dose of vaccine, approximately Day 56.

SECONDARY OUTCOMES:
GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group. | 1 month and 7 months after receipt of the 1st dose of vaccine.
GMT and frequency of 4-fold or greater increases in serum HAI antibody titers in each group. | 1 month and 7 months after receipt of the 1st dose of vaccine.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Keitel WA, Dekker CL, Mink C, Campbell JD, Edwards KM, Patel SM, Ho DY, Talbot HK, Guo K, Noah DL, Hill H. Safety and immunogenicity of inactivated, Vero cell culture-derived whole virus influenza A/H5N1 vaccine given alone or with aluminum hydroxide adjuvant in healthy adults. Vaccine. 2009 Nov 5;27(47):6642-8. doi: 10.1016/j.vaccine.2009.03.015. Epub 2009 Mar 25. PMID 19773098